CLINICAL TRIAL: NCT00554203
Title: Effect of Sulfasalazine on Endothelial Function
Brief Title: Sulfasalazine and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-22844
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sulfasalazine — sulfasalazine 2 grams daily for 6 weeks

SUMMARY:
Experimental studies suggest that systemic inflammation leads to endothelial dysfunction and atherosclerosis. This study will examine the effects of the anti-inflammatory drug sulfasalazine on endothelial function in patients with coronary artery disease. Subjects will be treated with sulfasalazine or to placebo for six weeks. After a two-week rest period, subjects will cross over to the alternative treatment. Endothelium-dependent flow-mediated dilation of the brachial artery will be studied before and after each drug. We hypothesize that anti-inflammatory therapy will reverse endothelial dysfunction in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease

Exclusion Criteria:

* G6PD deficiency defined by red blood cell G6PD activity assay
* Sulfa allergy
* Aspirin allergy
* Allergy to furosemide (lasix), hydrochlorthiazide, sulfonylureas, acetazolamide (Diamox) or other carbonic anhydrase inhibitors
* SGOT, SGPT, alkaline phosphatase, total bilirubin greater than 2 times the upper limit of normal
* WBC less than 4.0 or greater than 11.0 K/UL
* Platelet count less than 150 K or greater than 450K
* Hematocrit less than 30% 7
* Serum creatinine greater than 1.5 mg/dl
* Unstable angina or acute MI within 2 weeks
* Warfarin treatment
* Immunosuppressive treatment (methotrexate, cyclosporine, etc.)
* Digoxin treatment
* Phenytoin (Dilantin) treatment
* Methenamine (Mandelamine, Urex) treatment
* Probenecid or sulfinpyrazone (Anturane, Aprazone) treatment
* Porphyria
* Symptomatic GI obstruction
* GU obstruction (not including clinical evidence of benign prostatic hypertrophy)
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 6 weeks

SECONDARY OUTCOMES:
serum markers of inflammation | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Tabit CE, Holbrook M, Shenouda SM, Dohadwala MM, Widlansky ME, Frame AA, Kim BH, Duess MA, Kluge MA, Levit A, Keaney JF Jr, Vita JA, Hamburg NM. Effect of sulfasalazine on inflammation and endothelial function in patients with established coronary artery disease. Vasc Med. 2012 Apr;17(2):101-7. doi: 10.1177/1358863X12440117. PMID 22496207